CLINICAL TRIAL: NCT06237205
Title: Genome-Based Assessment of Niraparib (ZEJULA®) Efficacy in Advanced Solid TumorS With Homologous Recombination Deficiency (GAUSS)
Brief Title: Genome-Based Assessment of Niraparib (ZEJULA®) Efficacy in Advanced Solid TumorS With Homologous Recombination Deficiency
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Takeda (Industry); Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Lee, Soo Hyeon, Investigator, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAUSS
Record Dates: First submitted 2024-01-08; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Efficacy
MeSH Terms: interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niraparib (Experimental)
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — a highly selective PARP1 and PARP2 inhibitor

SUMMARY:
Investigational Products: Niraparib Period: 3 years after IRB/EC approval Indication: Adult patients with histologically confirmed and locally advanced, unresectable, or metastatic solid tumors having known or suspected deleterious mutations in genes involved in homologous recombination repair (HRR) or homologous recombination deficiency identified by whole genome sequencing

DETAILED DESCRIPTION:
Objectives:

1. Primary Objective

   - Antitumor activity defined as objective response at ≥ 8 weeks or stable disease (SD) at ≥ 16 weeks from the time of enrollment.
2. Secondary Objectives

   * Overall Survival (OS)
   * Progression-Free Survival (PFS)
   * Objective Response Rate (ORR) by RECIST v1.1
   * Duration of response (DOR)
   * Quality of life (QOL) assessed by EORTC-QLQ-C30
   * Adverse Event (AEs)
   * Exploratory biomarker analyses

ELIGIBILITY:
Inclusion Criteria:

1. Patient who agreed to participate in the KOSMOS-II master observation study.
2. 19 years of age or older on the day of signing informed consent.
3. Has a histologically- or cytologically-confirmed advanced (metastatic and/or unresectable) solid tumor.
4. Has either known or suspected deleterious mutations in at least 1 of the genes involved in HRR or centrally confirmed HRD based on whole-genome sequencing (WGS).
5. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
6. Has measurable disease per RECIST v1.1 as assessed by the local site investigator.
7. Female participants of reproductive potential must agree to use contraception during the treatment period and for at least 6 months after the last dose. Male participants must agree to use contraception during the treatment period and for 90 days plus 5 X half-life after last dose.
8. Has adequate organ function.
9. Willing to provide biopsies from the tumor at screening to the central laboratory

Exclusion Criteria:

1. Any previous exposure to PARP inhibitor
2. Any other active malignancy or diagnosis of another malignancy within 2 years before study enrollment
3. Has leptomeningeal metastases.
4. Active central nervous system (CNS) lesions.
5. Were resistant to prior platinum therapy (cisplatin, carboplatin, or oxaliplatin either as monotherapy or in combination) for advanced (metastatic and/or unresectable) solid tumor.
6. Any cytotoxic chemotherapy from a previous treatment regimen within 14 days.
7. Has received prior endocrine therapy as cancer treatment within 2 weeks prior to administration of study intervention.
8. Has received palliative radiotherapy encompassing >20% of the bone marrow within 1 week of the first dose of study treatment.
9. Has an active infection requiring systemic therapy.
10. Has hypertension that cannot be adequately controlled with medication.
11. Has active tuberculosis.
12. Has active infection such as hepatitis B, hepatitis C
13. Has a known history of Human Immunodeficiency Virus (HIV) infection.

15) Impairment of gastrointestinal function or gastrointestinal disorders 16) Is pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the screening visit through 6 months after the last dose of the Investigational product.

17) Patients who do not consent to adequate contraception throughout the study period.

18) Has a known hypersensitivity to the components of the investigational product or its analogs.

19) Since this drug contains lactose, patients with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.

20) Since this drug contains Yellow No. 4 (Tartrazine), patients with a history of hypersensitivity or allergy to this ingredient.

21) Medical, psychiatric, cognitive, or other conditions that may interfere with the ability of the subject to understand the subject information, provide the informed consent, follow the protocol process, or complete the clinical trial.

22) The investigator judges that it is not appropriate to participate in this study for else reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-02-27 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
objective response after 8 weeks | at 8 weeks after Cycle 1 Day 1(each cycle is 28 days)
  Antitumor activity defined as objective response after 8 weeks